CLINICAL TRIAL: NCT04827355
Title: Randomized Sham-Controlled Trial of the Reflux Band in Laryngopharyngeal Reflux (LPR)
Brief Title: Reflux Band in Laryngopharyngeal Reflux
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rena Yadlapati, Professor of Clinical Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201945; K23DK125266 (NIH)
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Laryngopharyngeal Reflux
Keywords: Proton Pump Inhibitor (PPI); Upper Esophageal Sphincter (UES) Compression Device
MeSH Terms: conditions — Laryngopharyngeal Reflux

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of two arms: control or experimental. Randomization will be 1:1 to control (sham, known not to provide intervention) and experimental (fit to manufacturer guidelines).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (Sham Comparator): Participants allocated to the control arm will be fit with the UES Compression Device at a pressure known not to provide intervention.
  Interventions: Device: Sham Device
- Experimental (Experimental): Participants allocated to the experimental arm will be fit with the UES Compression Device according to manufacturer guidelines.
  Interventions: Device: External Upper Esophageal Sphincter (UES) Compression Device

INTERVENTIONS:
Device: External Upper Esophageal Sphincter (UES) Compression Device — External Upper Esophageal Sphincter (UES) Compression Device fit to manufacturer guidelines.
  Other Names: Reflux Band; Reza Band
  Arms: Experimental
Device: Sham Device — External Upper Esophageal Sphincter (UES) Compression Device fit to pressure known not to provide treatment.
  Arms: Control

SUMMARY:
This 12 week biomarker targeted double blind randomized controlled trial (RCT) will enroll subjects with salivary pepsin positive laryngopharyngeal reflux (LPR) to assess efficacy of the external upper esophageal sphincter (UES) compression device, also known as the Reflux Band. Subjects will be randomized to one of two arms: control or experimental. Following the 8 week intervention period subjects in both arms will continue in a 4 week unblinded period. The primary hypothesis is that a significantly higher proportion of subjects in the experimental arm will meet the primary endpoint for symptom response, compared to subjects in the control arm.

DETAILED DESCRIPTION:
This study seeks to understand if the Reflux Band is an effective treatment for laryngopharyngeal reflux (LPR) in comparison to a sham device. LPR is a syndrome in which acid that is made in the stomach travels up the esophagus and into the throat, causing chronic symptoms including throat clearing, voice hoarseness, sore throat, etc. Participation in the study may or may not benefit you directly, and may result in new knowledge that may help others.

Participation in this study involves: 3 - 4 in person visits (2 of which are part of standard of care) ranging from 30 - 45 minutes each and 2 virtual visits, either by phone or video, each 15 minutes. Participants are assigned with a 50/50 chance (similar to a coin flip) via a computer generator to receive the Reflux Band or sham device (a device that will not provide you medical therapy) which they will wear around their neck nightly while sleeping (6+ hours) over a duration of 8 weeks. The Reflux Band, which has been cleared for use by the FDA, applies pressure to the outside of the neck at the cricoid cartilage, at the middle of the neck, and increases the internal pressure of the muscle separating the throat from the esophagus (upper esophageal sphincter). Participants will only wear the band while sleeping at night and remove in the morning upon waking. The in person visits will occur at one of these UCSD La Jolla locations: the Perlman Medical Office Gastroenterology clinic, the Center for Voice and Swallowing, Altman Clinical and Translational Research Institute (ACTRI) Clinic.

There is an optional 4 week extension at the end of this study in which the Reflux Band will be refit (if sham) to provide the manufacturer's specified pressure. This portion contains 1 virtual follow up during week 10 and an in person follow up during week 12, at which time study participation will conclude.

The most commonly expected risks of the study are skin reaction, discomfort, and difficulty sleeping. These were generally mild and short in duration. No serious risks were observed when the Reflux Band was worn around the neck in previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18-99, English or Spanish speaking
* ≥8 weeks of laryngeal symptoms (dysphonia, throat clearing, cough, globus, and/or sore throat)
* Current use of double daily dose acid suppression therapy (ex. omeprazole 40mg, omeprazole 20mg and famotidine 20mg)
* Laryngoscopic exam prior to screening with current symptoms
* At least 1 of the following:

  * Elevated reflux testing
  * Findings on upper endoscopy that are consistent with pathologic GERD
  * Fasting pepsin analysis result of ≥25 ng/mL within 4 months of enrollment (12 months if treatment plan has not changed) *testing allowed at enrollment if not previously obtained

Exclusion Criteria:

* Prior use of Reflux Band (UES Compression Device)
* Sino-pulmonary conditions (such as asthma, COPD, post-nasal drip, heavy voice use) as primary etiology of laryngeal symptoms as deemed by treating gastroenterologist and / or laryngologist
* Laryngeal mass or lesion on laryngoscopy
* Pregnant or breastfeeding
* Unable to consent in English or Spanish
* Imprisoned
* Patients with a prior foregut surgery
* Patients with a known achalasia diagnosis
* Inability to fast for 4 hours
* Active tobacco use
* Supplemental oxygen use
* Contraindication to UES Compression Device manufacturer guidelines:
* Patients with implants or implant parts that reside in the area where Reflux Band is applied: implanted pacemarker, implanted cardioverter defibrillator (ICD), vagus nerve stimulator (VNS), or other such devices implanted in the neck
* Patients diagnosed with glaucoma.
* Patients who had a malignancy of the neck, including neck surgery.
* Patients that may have an altered mental status including due to the use of sedative drugs or narcotics.
* Patients with carotid artery disease, uncontrolled thyroid disease, a history of cerebrovascular disease, or connective tissue disorder of Marfan's Syndrome or Ehlers-Danlos Syndrome
* Patients who use nocturnal NIV machines such as CPAP or BiPAP.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Measure response to the UES Compression Device in pepsin positive LPR. | 5 years
  Change in reflux symptom index score (primary outcome) between intervention versus sham arm will determine device efficacy.

SECONDARY OUTCOMES:
Measure pepsin response to the UES Compression Device in pepsin positive LPR. | 5 years
  Change in salivary pepsin concentration between pre and post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rena Yadlapati, MD, MSHS, Principal Investigator — UC San Diego Health
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Olson NR. Laryngopharyngeal manifestations of gastroesophageal reflux disease. Otolaryngol Clin North Am. 1991 Oct;24(5):1201-13. PMID 1754220
- [Background] Cohen SM, Pitman MJ, Noordzij JP, Courey M. Management of dysphonic patients by otolaryngologists. Otolaryngol Head Neck Surg. 2012 Aug;147(2):289-94. doi: 10.1177/0194599812440780. Epub 2012 Feb 24. PMID 22368039
- [Background] Ruiz R, Jeswani S, Andrews K, Rafii B, Paul BC, Branski RC, Amin MR. Hoarseness and laryngopharyngeal reflux: a survey of primary care physician practice patterns. JAMA Otolaryngol Head Neck Surg. 2014 Mar;140(3):192-6. doi: 10.1001/jamaoto.2013.6533. PMID 24481258
- [Background] Litvinov AV. [Method of tracheobronchial spraying of drugs in aerosols]. Vestn Khir Im I I Grek. 1976 Jan;116(1):100-1. No abstract available. Russian. PMID 1020172
- [Background] de Bortoli N, Nacci A, Savarino E, Martinucci I, Bellini M, Fattori B, Ceccarelli L, Costa F, Mumolo MG, Ricchiuti A, Savarino V, Berrettini S, Marchi S. How many cases of laryngopharyngeal reflux suspected by laryngoscopy are gastroesophageal reflux disease-related? World J Gastroenterol. 2012 Aug 28;18(32):4363-70. doi: 10.3748/wjg.v18.i32.4363. PMID 22969200
- [Result] Shaker R, Babaei A, Naini SR. Prevention of esophagopharyngeal reflux by augmenting the upper esophageal sphincter pressure barrier. Laryngoscope. 2014 Oct;124(10):2268-74. doi: 10.1002/lary.24735. Epub 2014 Jun 27. PMID 24782387
- [Result] Slivers SL, Vaezi MF, Vakil MB, et al. Prospective study of upper esophageal sphincter assist device for treating extraesophageal reflux. Otolaryngol Open J. 2016; 2(1): 31-38. doi: 10.17140/OTLOJ-2-109
- [Result] Yadlapati R, Craft J, Adkins CJ, Pandolfino JE. The Upper Esophageal Sphincter Assist Device Is Associated With Symptom Response in Reflux-Associated Laryngeal Symptoms. Clin Gastroenterol Hepatol. 2018 Oct;16(10):1670-1672. doi: 10.1016/j.cgh.2018.01.031. Epub 2018 Jan 31. PMID 29408585
- [Derived] Yadlapati R, Robles L, Clarke MK, Low EE, Walsh E, Krause AJ, Kaizer A. Randomized Controlled Trial of Upper Esophageal Sphincter Assist Device in Laryngopharyngeal Reflux Disease. Clin Gastroenterol Hepatol. 2025 Dec 22:S1542-3565(25)01062-6. doi: 10.1016/j.cgh.2025.12.015. Online ahead of print. PMID 41443523

DOCUMENTS (1):
  • Informed Consent Form (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT04827355/ICF_002.pdf